CLINICAL TRIAL: NCT03226249
Title: Phase II Study of PET-Directed Frontline Therapy With Pembrolizumab and AVD for Patients With Classical Hodgkin Lymphoma
Brief Title: PET-Directed Therapy With Pembrolizumab and Combination Chemotherapy in Treating Patients With Previously Untreated Classical Hodgkin Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Jane N. Winter, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 16H08; NU 16H08 (Other: Northwestern University); P30CA060553 (NIH); NCI-2017-00457 (Other: CTRP (Clinical Trial Reporting Program)); STU00203707 (Other: Northwestern University IRB#)
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Results first posted 2020-07-15 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Classical Hodgkin Lymphoma; Lymphocyte-Depleted Classical Hodgkin Lymphoma; Lymphocyte-Rich Classical Hodgkin Lymphoma; Mixed Cellularity Classical Hodgkin Lymphoma; Nodular Sclerosis Classical Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Dacarbazine; Doxorubicin; Fluorodeoxyglucose F18; pembrolizumab; Magnetic Resonance Spectroscopy; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (FDG-PET/CT, pembrolizumab, chemotherapy) (Experimental): See Detailed Description
  Interventions: Procedure: Computed Tomography; Drug: Dacarbazine; Drug: Doxorubicin Hydrochloride; Radiation: Fludeoxyglucose F-18; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Procedure: Positron Emission Tomography; Drug: Vinblastine Sulfate

INTERVENTIONS:
Procedure: Computed Tomography — Undergo FDG-PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Drug: Dacarbazine — Given IV
  Other Names: 4-(Dimethyltriazeno)imidazole-5-carboxamide; 5-(Dimethyltriazeno)imidazole-4-carboxamide; Asercit; Biocarbazine; Dacarbazina; Dacarbazina Almirall; Dacarbazine - DTIC; Dacatic; Dakarbazin; Deticene; Detimedac; DIC; Dimethyl (triazeno) imidazolecarboxamide; Dimethyl Triazeno Imidazol Carboxamide; Dimethyl Triazeno Imidazole Carboxamide; dimethyl-triazeno-imidazole carboxamide; Dimethyl-triazeno-imidazole-carboximide; DTIC; DTIC-Dome; Fauldetic; Imidazole Carboxamide; Imidazole Carboxamide Dimethyltriazeno; WR-139007
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Radiation: Fludeoxyglucose F-18 — Undergo FDG-PET/CT
  Other Names: 18FDG; FDG; fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Procedure: Positron Emission Tomography — Undergo FDG-PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Drug: Vinblastine Sulfate — Given IV
  Other Names: 29060 LE; 29060-LE; Exal; Velban; Velbe; Velsar; VINCALEUKOBLASTINE

SUMMARY:
The purpose of this research study is to evaluate a new drug pembrolizumab in combination with chemotherapy, for the treatment of newly diagnosed Hodgkin lymphoma. The chemotherapy regimen is called AVD and includes three drugs: adriamycin, vinblastin, dacarbazine. Pembrolizumab is currently FDA approved for the treatment of some patients with melanoma, lung cancer and head and neck cancer, but has not yet been approved for the treatment of Hodgkins Lymphoma. The AVD regimen of chemotherapy is currently FDA approved for the treatment of newly diagnosed Hodgkin lymphoma, but has not yet been investigated in combination with pembrolizumab for this disease. For patients who have a new diagnosis of Hodgkins Lymphoma, multi-agent chemotherapy is recommended. Also, for patients who do not have a complete response to chemotherapy (meaning there is still evidence of disease on PET scans performed at the end of treatment), radiation is sometimes recommended. Furthermore, the rare patient who relapses after chemotherapy requires treatment with high dose chemotherapy and a transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the percent of patients who achieve a complete response (CR) to single-agent pembrolizumab induction, among patients with classical Hodgkin lymphoma (cHL) using Lugano 2014 criteria., as measured at PET #2.

SECONDARY OBJECTIVES:

I. Assess the safety and tolerability of pembrolizumab in combination with chemotherapy in the frontline setting.

II. Determine the three-year progression free survival (PFS) and overall survival (OS) for patients < 60 with early non-bulky disease, and elderly patients (all stages) treated with pembrolizumab with doxorubicin hydrochloride (Adriamycin), (bleomycin), vinblastine sulfate, dacarbazine (A[B]VD) in the frontline treatment of patients with cHL.

III. Determine the extent of fludeoxyglucose F-18 (FDG) uptake, using a semi-quantitative approach (e.g., Deauville score), after pembrolizumab induction, and after subsequent chemotherapy.

TERTIARY OBJECTIVES:

I. To characterize PD-1 pathway specific expression and correlate with response.

II. To characterize serum biomarkers of immune and inflammatory response during treatment.

III. To characterize levels of soluble PD-L1 related to treatment with pembrolizumab.

IV. To characterize T-lymphocyte subset changes to treatment with pembrolizumab.

V. To investigate the prevalence and clinical correlation of chromosome 9p24.1 alterations for this population.

OUTLINE:

INITIATION: Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients also undergo FDG-PET/computed tomography (CT) scans before the start of pembrolizumab and after 3 courses.

AVD: Within 21 days after final dose of pembrolizumab, patients receive doxorubicin hydrochloride IV, vinblastine sulfate IV, and dacarbazine IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo a final FDG-PET/CT scan on day 117-120 or 26-29 of course 2. Patients with stage I/II disease with a CR continue treatment for up to 2 courses. Patients with stage III/IV disease with a CR or age >= 60 with stage III/IV disease with any response continue treatment for up to 4 courses.

CONSOLIDATION: Patients age >= 60 with stage III/IV disease who received < 6 courses of AVD or patients age >= 60 with DV 4-5 on FDG-PECT/CT scan receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 17 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of classical Hodgkin lymphoma including nodular sclerosis, mixed cellularity, lymphocytic-rich, and lymphocyte depleted subtypes by the 4th edition of the World Health Organization (WHO) Classification of Tumors of Hematopoietic and Lymphoid Tissues published in 2008 (nodular lymphocyte-predominant Hodgkin lymphoma [NLPHL] excluded)
* Patients must have measurable disease by the Lugano criteria
* Patients must have previously untreated disease (except for one week or less of corticosteroids)
* Patients must exhibit a/an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Patients may have any stage and any International Prognostic Score (IPS)
* Patients must have adequate organ and bone marrow function within 14 days prior to registration, as defined below:
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcl
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal (ULN)
* Creatinine within normal institutional limits
* Platelet transfusions are acceptable prior to treatment to achieve the above numbers, however growth factors are not allowed within 14 days of registration
* Females of child-bearing potential (FOCBP) and males must agree to avoid becoming pregnant, or impregnating a partner, respectively, by complying with any of the approved contraception techniques prior to registration, for the duration of study participation, and for 120 days following completion of therapy; abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject; should a female patient become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy
* Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)

  * FOCBP must have a negative pregnancy test within 7 days prior to registration on study; NOTE: a negative pregnancy test is also required within 3 days prior to first dose of pembrolizumab and therefore may need to be repeated if screening test is more than 3 days prior to first dose
  * Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

* Patients are not eligible who have had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to registration or who have not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * NOTE: Subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * NOTE: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Patients who have a diagnosis of immunodeficiency or are receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to registration are not eligible
* Patients who have a known history of active TB (bacillus tuberculosis) are not eligible
* Patients must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
* Patients who have a known additional malignancy that is progressing or requires active treatment are not eligible

  * NOTE: Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Patients who have known active central nervous system (CNS) metastases and/or carcinomatous meningitis are not eligible

  * NOTE: Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to registration; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* Patients who have active autoimmune disease that has required systemic treatment in the past 2 years are not eligible (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs)

  * NOTE: Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Patients who have known history of, or any evidence of active, non-infectious pneumonitis are not eligible
* Patients who have an active infection requiring systemic therapy are not eligible, except for uncomplicated urinary tract infections
* Patients are not eligible who have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject?s participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Patients who have known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial are not eligible
* Patients may not be pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, from registration through 120 days after the last dose of trial treatment
* Patients who have received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent are not eligible
* Patients who have a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies) are not eligible
* Patients who have active hepatitis B (e.g., hepatitis B virus surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis c virus [HCV] ribonucleic acid [RNA] [qualitative] is detected) are not eligible
* Patients who received a live vaccine within 30 days of planned start of study therapy are not eligible; examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, bacillus Calmette-Guerin (BCG), and typhoid vaccine

  * NOTE: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2024-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Winter, M.D., Principal Investigator — Northwestern University
Locations (4):
- United States (4):
  - Stanford Cancer Institute, Stanford, California
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rutgers Cancer Institute, New Brunswick, New Jersey

REFERENCES:
- [Derived] Kreuzberger N, Goldkuhle M, von Tresckow B, Kobe C, Sickinger MT, Monsef I, Skoetz N. Positron emission tomography-adapted therapy for first-line treatment in adults with Hodgkin lymphoma. Cochrane Database Syst Rev. 2025 Mar 26;3(3):CD010533. doi: 10.1002/14651858.CD010533.pub3. PMID 40135712
- [Derived] Allen PB, Lu X, Chen Q, O'Shea K, Chmiel JS, Slonim LB, Sukhanova M, Savas H, Evens AM, Advani R, Pro B, Karmali R, Palmer B, Bayer RA, Eisner RM, Mou E, Dillehay G, Gordon LI, Winter JN. Sequential pembrolizumab and AVD are highly effective at any PD-L1 expression level in untreated Hodgkin lymphoma. Blood Adv. 2023 Jun 27;7(12):2670-2676. doi: 10.1182/bloodadvances.2022008116. PMID 36083129
- [Derived] Allen PB, Savas H, Evens AM, Advani RH, Palmer B, Pro B, Karmali R, Mou E, Bearden J, Dillehay G, Bayer RA, Eisner RM, Chmiel JS, O'Shea K, Gordon LI, Winter JN. Pembrolizumab followed by AVD in untreated early unfavorable and advanced-stage classical Hodgkin lymphoma. Blood. 2021 Mar 11;137(10):1318-1326. doi: 10.1182/blood.2020007400. PMID 32992341

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to accrual on September 6th, 2017 with an accrual goal of 30 patients. The first patient was enrolled onto the study and started treatment on November 9th, 2017. The study closed permanently to further enrollment of participants on March,12th 2019 as the accrual goal was met.
Groups:
- Treatment: Pembrolizumab and AVD Chemotherapy Guided by PET-CT: All patients get 3 cycles (21-days each) of pembrolizumab (PEM) induction, then a PET-CT (PET#2). PET#2 required for primary endpoint analysis. Patients evaluable for response assessment if they had at least one dose of PEM.
  After, all patients get 2 cycles (28-days each) of AVD (doxorubicin, vinblastine, dacarbazine), followed by an interim PET-CT (PET#3) for response analysis.
  Depending on age, stage, and PET#3 results per Deauville (DV) Score, patients get additional 2-4 cycles of AVD, or AVD and escBEACOPP (escalated bleomycin, etoposide, doxorubicin, cyclophosphamide, vincristine, procarbazine, prednisone) + radiotherapy (RT). Then, patients will have a PET-CT (PET#4) or a CT (CT if Stage I/II disease and negative for PET#3).
  Patients under 60 go to survival follow-up. Patients over 60 go to survival follow-up or 1-2 years of PEM consolidation based on bulky vs non bulky disease, results of the PET#3, and the number of AVD cycles received.
  See schema for details.
Period: PEM Induction Cycles 1-3, and PET#2
Arm/Group | Treatment: Pembrolizumab and AVD Chemotherapy Guided by PET-CT
Started | 30
PEM Cycle 1 | 30
PEM Cycle 2 | 30
PEM Cycle 3 | 30
PET#2 | 30
Completed | 30
Not Completed | 0
Period: 2 Cycles of AVD + PET#3
Arm/Group | Treatment: Pembrolizumab and AVD Chemotherapy Guided by PET-CT
Started | 30
AVD Cycle 1 | 30
AVD Cycle 2 | 30
PET#3 | 30
Completed | 30
Not Completed | 0
Period: 2-4 Cycles of AVD +/- Chemo & RT, PET#4
Arm/Group | Treatment: Pembrolizumab and AVD Chemotherapy Guided by PET-CT
Started | 30
2-4 Cycles of AVD +/- Chemo & RT | 29
PET#4 | 29
Completed | 29
Not Completed | 1
Not completed — Transferred to another state | 1
Period: PEM Consolidation (1-2 Years)
Arm/Group | Treatment: Pembrolizumab and AVD Chemotherapy Guided by PET-CT
Started | 29
Completed | 0
Not Completed | 29
Not completed — Per Protocol not eligible | 29
Period: Survival Follow-up
Arm/Group | Treatment: Pembrolizumab and AVD Chemotherapy Guided by PET-CT
Started | 30 (All patients that are treated with one dose of study drug go into follow-up.)
Completed | 0
Not Completed | 30
Not completed — Patients still in follow-up. | 30

BASELINE CHARACTERISTICS:
Arm/Group | Treatment: Pembrolizumab and AVD Chemotherapy Guided by PET-CT
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 25
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
Disease Stage [Count of Participants; unit: Participants] — Low stage number = less disease involvement. I: single lymph node (LN) region or lymphoid structure. II: two or more LN regions or LN structures on the same side of the diaphragm. III: LN regions or lymphoid structures on both sides of the diaphragm. IV: Diffuse or dissemination of one or more extranodal organs or tissue beyond, with or without associated LN involvement. *A/B to indicate the absence (A) or presence (B) of the systemic symptoms of significant unexplained fever, night sweats, or unexplained weight loss exceeding 10% of body weight during 6 months prior to diagnosis.
  Participants
    IIa | 6
    IIb | 6
    IIIa | 4
    IIIb | 1
    IVa | 6
    IVb | 7
Bulky vs Non-Bulky Disease [Count of Participants; unit: Participants] — Per Protocol, bulky disease is a mass >10 cm.
  Participants
    Yes | 14
    No | 16

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) With Pembrolizumab Treatment Alone
Description: To assess the primary objective of response rate following PET #2 performed after 3 doses of pembrolizumab. PET response will be assessed using the Lugano Criteria (2014) which recommends the 5 point Deauville score for assessing response. The Deauville five-point scale is an internationally-recommended scale for routine clinical reporting and clinical trials using FDG PET-CT in the initial staging and assessment of treatment response in Hodgkin lymphoma (HL). Patients with a Deauville score of 1-3 will be considered a complete response.
  Deauville criteria is defined as follows:
  1. No residual uptake
  2. Slight uptake, but below blood pool (mediastinum)
  3. Uptake above mediastinum, but below or equal to uptake in the liver
  4. Uptake slightly to moderately higher than liver
  5. Markedly increased uptake or any new lesions
  Patients will be evaluable for response assessment if they have received at least one dose of pembrolizumab.
Time Frame: After 3 cycles of pembrolizumab (1 cycle = 21 days)
Measure: Number; unit: percentage of participants
Arm/Group | Treatment: Pembrolizumab and AVD Chemotherapy Guided by PET-CT
Number analyzed (Participants) | 30
percentage of participants | 37

2. Secondary Outcome: Incidence of Adverse Events
Description: To assess safety and tolerability, all adverse events will be summarized in terms of type, grade, timing and attribution to treatment and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 (NCI-CTCAE version 4.03).
Time Frame: Up to 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Progression Free Survival (PFS) for Patients <60
Description: PFS for patients <60 will be measured.
Time Frame: Up to 2 years
Reporting Status: Not Posted

4. Secondary Outcome: PFS for Elderly Patients
Description: PFS for elderly patients will be measured.
Time Frame: Up to 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Overall Survival (OS) for Patients <60
Description: OS for patients <60 will be evaluated.
Time Frame: Up to 2 years
Reporting Status: Not Posted

6. Secondary Outcome: OS for Elderly Patients
Description: OS for elderly patients will be evaluated.
Time Frame: Up to 2 years
Reporting Status: Not Posted

7. Secondary Outcome: FDG Uptake
Description: Evaluate the extent of FDG uptake by assessing PET scans to determine a Deauville score.
Time Frame: Up to 4 weeks after last dose of chemotherapy
Reporting Status: Not Posted

8. Post Hoc Outcome: Progression Free Survival (PFS) at Treatment Completion
Description: PFS is defined as the number of patients that are progression/relapse free at the time of treatment completion (3 cycles of pembrolizumab and up to 6 cycles of AVD).
  Progressive or relapse disease is defined as of the following:
  Appearance of any new lesion more than 1.5 cm in any axis during treatment, even if other lesions are decreasing in size.
  At least a 50% increased from nadir in the sum of the product of the diameter (SPD) of any previously involved nodes, or in a single involved node, or the size of other lesions (e.g., splenic or hepatic nodules). To be considered progressive disease, a lymph node with a diameter of the short axis of less than 1.0 cm must increase by at least 50% and to a size of more than 1.5 x 1.5 cm or more than 1.5 cm in the long axis.
  At least a 50% increase in the longest diameter of any single previously identified node more than 1.0 cm in its short axis.
  Lymphoma confirmed by repeat biopsy.
Time Frame: At completion of treatment with 3 cycles of pembrolizumab (21 day cycles) and up to 6 cycles of AVD (28 days cycles)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: Pembrolizumab and AVD Chemotherapy Guided by PET-CT
Number analyzed (Participants) | 30
Participants | 30

9. Post Hoc Outcome: Overall Survival at Treatment Completion
Description: Overall survival will be defined as the number of patients that are alive at the time of treatment completion (3 cycles of pembrolizumab and 2-6 cycles of AVD)
Time Frame: At completion of treatment with 3 cycles of pembrolizumab (21 day cycles) and up to 6 cycles of AVD (28 days cycles)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: Pembrolizumab and AVD Chemotherapy Guided by PET-CT
Number analyzed (Participants) | 30
Participants | 30

ADVERSE EVENTS:
Time Frame: Up to 3 cycles of pembrolizumab (21 day cycles), and up to 6 cycles of AVD (28 day cycles), or approximately 33 weeks.
Description: Adverse event data shown below includes all events collected and available up until March 23rd 2020 for the study. Data collected includes the highest grade of the event experienced for each participant, and thus includes some serious adverse event data. Adverse event data
Arm/Group | Treatment: Pembrolizumab and AVD Chemotherapy Guided by PET-CT
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 6/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment: Pembrolizumab and AVD Chemotherapy Guided by PET-CT (N=30)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) — The participant also experienced increased aspartate aminotransferase, alanine aminotransferase, and alkaline phosphatase at the time of the event.
Pericarditis (Cardiac disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment: Pembrolizumab and AVD Chemotherapy Guided by PET-CT (N=30)
Anemia (Blood and lymphatic system disorders) | 22
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 4
Palpitations (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 0
Sinus tachycardia (Cardiac disorders) | 3
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 2
Hearing impaired (Ear and labyrinth disorders) | 0
Tinnitus (Ear and labyrinth disorders) | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Hyperparathyroidism (Endocrine disorders) | 0
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Blurred vision (Eye disorders) | 2
Cataract (Eye disorders) | 0
Conjunctivitis (Eye disorders) | 1
Dry eye (Eye disorders) | 2
Eye disorders - Other, specify (Eye disorders) | 0
Watering eyes (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 0
Abdominal pain (Gastrointestinal disorders) | 6
Anal hemorrhage (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 20
Diarrhea (Gastrointestinal disorders) | 9
Dyspepsia (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 5
Hemorrhoids (Gastrointestinal disorders) | 0
Mucositis oral (Gastrointestinal disorders) | 15
Nausea (Gastrointestinal disorders) | 23
Oral pain (Gastrointestinal disorders) | 3
Rectal hemorrhage (Gastrointestinal disorders) | 3
Rectal pain (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Chills (General disorders) | 3
Edema limbs (General disorders) | 3
Fatigue (General disorders) | 20
Fever (General disorders) | 6
Flu like symptoms (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 6
Infusion related reaction (General disorders) | 5
Localized edema (General disorders) | 1
Malaise (General disorders) | 7
Non-cardiac chest pain (General disorders) | 7
Pain (General disorders) | 7
Allergic reaction (Immune system disorders) | 3
Immune system disorders - Other, specify (Immune system disorders) | 0
Gum infection (Infections and infestations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 0
Mucosal infection (Infections and infestations) | 1
Papulopustular rash (Infections and infestations) | 0
Peripheral nerve infection (Infections and infestations) | 0
Pharyngitis (Infections and infestations) | 2
Rash pustular (Infections and infestations) | 1
Rhinitis infective (Infections and infestations) | 2
Sepsis (Infections and infestations) | 0
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 3
Small intestine infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 2
Bruising (Injury, poisoning and procedural complications) | 3
Burn (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 2
Activated partial thromboplastin time prolonged (Investigations) | 0
Alanine aminotransferase increased (Investigations) | 11
Alkaline phosphatase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 12
Blood bilirubin increased (Investigations) | 3
Creatinine increased (Investigations) | 2
INR increased (Investigations) | 1
Investigations - Other, specify (Investigations) | 0
Lymphocyte count decreased (Investigations) | 18
Neutrophil count decreased (Investigations) | 28
Platelet count decreased (Investigations) | 2
Weight gain (Investigations) | 3
Weight loss (Investigations) | 4
White blood cell decreased (Investigations) | 28
Anorexia (Metabolism and nutrition disorders) | 10
Dehydration (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 23
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 5
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 11
Hypocalcemia (Metabolism and nutrition disorders) | 9
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 11
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 6
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Myositis (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0
Ataxia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
Facial nerve disorder (Nervous system disorders) | 0
Headache (Nervous system disorders) | 10
Memory impairment (Nervous system disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 0
Paresthesia (Nervous system disorders) | 2
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 8
Presyncope (Nervous system disorders) | 1
Sinus pain (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 6
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 8
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2
Urinary frequency (Renal and urinary disorders) | 3
Urinary retention (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 3
Urinary urgency (Renal and urinary disorders) | 1
Breast pain (Reproductive system and breast disorders) | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1
Irregular menstruation (Reproductive system and breast disorders) | 4
Ovulation pain (Reproductive system and breast disorders) | 0
Pelvic pain (Reproductive system and breast disorders) | 2
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0
Vaginal discharge (Reproductive system and breast disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7
Pharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 10
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 10
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 8
Rash acneiform (Skin and subcutaneous tissue disorders) | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 5
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0
Hot flashes (Vascular disorders) | 4
Hypertension (Vascular disorders) | 19
Hypotension (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 2
Vascular disorders - Other, specify (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT03226249/Prot_SAP_000.pdf